CLINICAL TRIAL: NCT00525356
Title: INvestigation of STEnt Grafts in Patients With Type B Aortic Dissection
Brief Title: INSTEAD Trial: INvestigation of STEnt Grafts in Patients With Type B Aortic Dissection
Acronym: INSTEAD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Organization: Medtronic Cardiovascular (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INSTEAD trial
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2007-09

CONDITIONS: Aortic Diseases
Keywords: Aorta; Dissection; Thoracic
MeSH Terms: conditions — Aortic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Active Comparator): Anti-hypertensive medical treatment
  Interventions: Device: Medtronic Talent Stent-Graft-System

INTERVENTIONS:
Device: Medtronic Talent Stent-Graft-System
  Other Names: Endograft

SUMMARY:
The objective of this study is to compare treatment with an endograft prothesis versus antihypertensive treatment in patients with a dissection of the thoracic aorta.

DETAILED DESCRIPTION:
Patients older than 18 years with type B aortic dissection as diagnosed by computed tomography or magnetic resonance angiography are randomized to either a thoracic aortic endoprosthesis and antihypertensive treatment, called "stent grafting," or a tailored antihypertensive treatment, called "medical treatment."

Only patients in a clinically stable condition and without spontaneous thrombosis of the false lumen after 14 days of the index dissection are considered eligible for study inclusion.

Primary outcome measure is all-cause mortality. Secondary outcome variables include conversion to stent and/or surgery, induced thrombosis of the false lumen, cardiovascular morbidity, aortic expansion (>5 mm/y of maximum diameter including true and false lumina), quality of life, and length of intensive care unit and hospital stay. The study design calls for 136 patients to be randomized and monitored for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* No contraindication for an anesthetic procedure with intubation
* Type B aortic dissection that occurred 2-52 weeks before randomization
* Diameter of the targeted aortic segment ≤6 cm
* Aortic kinking <75°
* The subject or legal guardian understands the nature of the study and agrees to its provisions on a written informed consent form
* Availability for the appropriate follow-up visits during the follow-up period
* Capability to follow all study requirements

Exclusion Criteria:

* Pregnant woman
* Thrombocytopenia or ongoing anticoagulation therapy
* Renal failure and/or creatinine >2.4 mg%
* Complete thrombosis of the false lumen
* Ongoing infection
* Cancer is likely to cause death within 1 year
* Enrolment in another clinical study
* Unwillingness to cooperate with study procedures or follow-up visits

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2002-02; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
all-cause mortality | 1 year

SECONDARY OUTCOMES:
thrombosis of the false lumen, cardiovascular morbidity, degree of aortic expansion, length of intensive care and hospital stay, and quantitative assessment of single or combination antihypertensive drug therapy. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: C A Nienaber, MD, FESC, FACC, Principal Investigator — Division of Cardiology and Internal Medicine Department, Rostock University, Germany.
Locations (1):
- Medtronic Bakken Research Center, Maastricht, Netherlands

REFERENCES:
- [Background] Nienaber CA, Zannetti S, Barbieri B, Kische S, Schareck W, Rehders TC; INSTEAD study collaborators. INvestigation of STEnt grafts in patients with type B Aortic Dissection: design of the INSTEAD trial--a prospective, multicenter, European randomized trial. Am Heart J. 2005 Apr;149(4):592-9. doi: 10.1016/j.ahj.2004.05.060. PMID 15990739
- [Background] Nienaber CA, Rousseau H, Eggebrecht H, Kische S, Fattori R, Rehders TC, Kundt G, Scheinert D, Czerny M, Kleinfeldt T, Zipfel B, Labrousse L, Ince H; INSTEAD Trial. Randomized comparison of strategies for type B aortic dissection: the INvestigation of STEnt Grafts in Aortic Dissection (INSTEAD) trial. Circulation. 2009 Dec 22;120(25):2519-28. doi: 10.1161/CIRCULATIONAHA.109.886408. Epub 2009 Dec 7. PMID 19996018